CLINICAL TRIAL: NCT05046717
Title: Improvement of Immunologic and Molecular Techniques for the Diagnosis and Follow-up of Patients With Thrombotic Thrombocytopenic Purpura: a Collaborative Study Proposal of the Spanish Apheresis Group (GEA) in Collaboration With the Spanish Foundation of Hematology and Hemotherapy (FEHH)
Brief Title: Improvement of Immunologic and Molecular Techniques for the Diagnosis and Follow-up of Patients With Thrombotic Thrombocytopenic Purpura
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación Española de Hematología y Hemoterapía (Other)
Responsible Party: Sponsor
Other Study IDs: INSPIRER
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — • Patients between 0 to 99 years old at the time of screeningwith confirmed thrombotic microangiopathy (TMA) based on citrated blood samples meeting both of the following criteria:
  * Thrombocytopenia [drop in platelet count ≥50% or platelet count < 100x109/L and
  * Microangiopathic haemolytic anaemia (elevation of lactate dehydrogenase (LDH) >2-fold or by presence or increase of schistocytes in peripheral blood smear)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ADAMTS13 Activity Assays — In this study the measurement of ADAMTS13 activity will be assessed with three different commercial kits:
  1. HemosIL AcuStar ADAMTS13 Activity Assay (Instrumentation Laboratory, Bedford, Massachusetts, United States)
  2. ELISA, DG-EIA ADAMTS13 Activity (Diagnostic Grifols®, Spain)
  3. FRETS-VWF73 for ADAMTS13 Activity Assay
  Three kits will be used with all patients.

SUMMARY:
The lack of ADAMTS13 is the only biological marker that is specific for aTTP diagnosis8 and the assessment of ADAMTS13 is of clinical importance because it is essential for the rapid differential diagnosis between aTTP and other TMA. Furthermore, monitoring of ADAMTS13 activity is useful to ensure biological remission (ADAMTS13 levels > 10%) as well as predicting relapses.

Due to the high mortality rate of aTTP, treatment should be started as soon as the disease is suspected, sometimes even before confirmation with the ADAMTS13 test results. This situation may lead to misdiagnose some patients and leave them without the appropriate treatment. In conclusion, ADAMTS13 activity assay is crucial for an early diagnosis and optimal management of acute aTTP and any delay in ADAMTS13 results will have a negative impact on the diagnosis, treatment and prognosis of the patient.

There are currently 2 techniques available for the ADAMTS13 activity determination, the fluorescence resonance energy transfer (FRET) and the Technozym chromogenic enzyme-linked immunosorbent assay (ELISA). Both are considered reference methods but they require considerable skill because they are highly manual and this increases the risk of error. Furthermore, these methods are time-consuming, not widely available and, in case of the ELISA method, it requires a new calibration at each run. The inter-laboratory variability is also a challenge and therefore a validation and/or interpretation method could be needed.

Recently, a new and first fully automated HemosIL AcuStar ADAMTS13 Activity assay (Instrumentation Laboratory, Bedford, Massachusetts, United States) has been developed. HemosIL AcuStar ADAMTS13 Activity assay is a two steps chemiluminescent immunoassay (CLIA) with an analytical time of 33 minutes for the quantitative measurement of ADAMTS13 activity in human-citrated plasma on the ACL AcuStar analyser. The immunoassay uses the GST-VWF73 substrate in combination with magnetic particles for rapid separation and chemiluminescence technology detection. The ADAMTS13 present in the plasma sample cleavages the GST-VWF73 substrate and the detection of the generated fragments is based upon an isoluminol-labelled monoclonal antibody that specifically reacts with the cleaved peptide. The emitted light is proportional to the ADAMTS13 activity in the sample.

This new ADAMTS13 assay method has been compared with the other two available techniques in two different studies. First, Favresse et al. published the results of the comparison between Technozym activity ELISA assay and the new HemosIL AcuStar chemiluminescent assay. On the other hand, Valsecchi et al. have recently published the results of validation of this new technique in comparison with ELISA and FRETS in 176 samples. Both studies conclude that the new chemiluminescent ADAMTS13 activity assay showed a good correlation and excellent clinical performance for the diagnosis of severe ADAMTS13 deficiency with the FRETS-VWF73 assay and a commercial ELISA when considering only ADAMTS13 activity values below 10% (the internationally accepted cut-off for a diagnosis of severe ADAMTS13 deficiency typical of aTTP). Finally, Stratmann et al. have just published another study comparing the HemosIL AcuStar chemiluminescent assay with two commercially available ADAMTS13 assay kits using 24 paired test samples derived from 10 consecutively recruited patients13 and their results corroborate the previously published data suggesting that the AcuStar assay could be a valuable and accurate tool for ADAMTS13 activity testing and aTTP diagnostic.

In this context, a unique opportunity to validate this new technique is generated, both retrospectively with our already available data from frozen samples and also in the context of a large prospective study. This will be the first study worldwide testing HemosIL AcuStar method in real clinical practice aTTP population (Spanish and Portuguese aTTP populations) with the aim to standardize the diagnosis and follow-up methodology for the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed thrombotic microangiopathy (TMA) based on citrated blood samples meeting both of the following criteria:

  * Thrombocytopenia [drop in platelet count ≥50% or platelet count < 100x109/L and
  * Microangiopathic haemolytic anaemia (elevation of lactate dehydrogenase (LDH) >2- fold or by presence or increase of schistocytes in peripheral blood smear)
* Patients that voluntarily sign informed consent. For subjects unable to provide consent, a fully recognized medical proxy may be used according to local laws.
* Patients between 0 to 99 years old at the time of screening.

Exclusion Criteria:

-

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be all consecutive patients who meet the following inclusion criteria and none of the following exclusion criteria until reaching the number of patients determined for the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of a new diagnostic test and standard test | At diagnosis of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Correlation of a new diagnostic test, HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS in the measurement of activity and antibody of ADAMTS13 in IU/mL
Correlation of a new diagnostic test and standard test | At follow up (10 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Correlation of a new diagnostic test, HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS in the measurement of activity and antibody of ADAMTS13 in IU/mL
Correlation of a new diagnostic test and standard test | At follow up (30 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Correlation of a new diagnostic test, HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS in the measurement of activity and antibody of ADAMTS13 in IU/mL
Correlation of a new diagnostic test and standard test | At follow up (60 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Correlation of a new diagnostic test, HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS in the measurement of activity and antibody of ADAMTS13 in IU/mL
Correlation of a new diagnostic test and standard test | At follow up (90 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Correlation of a new diagnostic test, HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS in the measurement of activity and antibody of ADAMTS13 in IU/mL
Correlation of a new diagnostic test and standard test | At follow up (180 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Correlation of a new diagnostic test, HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS in the measurement of activity and antibody of ADAMTS13 in IU/mL
Correlation of a new diagnostic test and standard test | At follow up (365 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Correlation of a new diagnostic test, HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS in the measurement of activity and antibody of ADAMTS13 in IU/mL

SECONDARY OUTCOMES:
Concordance of classification of aTTP | At diagnosis of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the concordance of classification of aTTP patients at diagnosis based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Concordance of classification of aTTP | At follow up (10 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the concordance of classification of aTTP patients based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Concordance of classification of aTTP | At follow up (30 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the concordance of classification of aTTP patients based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Concordance of classification of aTTP | At follow up (60 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the concordance of classification of aTTP patients based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Concordance of classification of aTTP | At follow up (90 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the concordance of classification of aTTP patients based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Concordance of classification of aTTP | At follow up (180 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the concordance of classification of aTTP patients based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Concordance of classification of aTTP | At follow up (365 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the concordance of classification of aTTP patients based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Sensitivity and specificity of classification of aTTP | At diagnosis of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the sensitivity and specificity of classification of aTTP patients visits based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Sensitivity and specificity of classification of aTTP | At follow up (10 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the sensitivity and specificity of classification of aTTP patients visits based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Sensitivity and specificity of classification of aTTP | At follow up (30 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the sensitivity and specificity of classification of aTTP patients visits based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Sensitivity and specificity of classification of aTTP | At follow up (60 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the sensitivity and specificity of classification of aTTP patients visits based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Sensitivity and specificity of classification of aTTP | At follow up (90 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the sensitivity and specificity of classification of aTTP patients visits based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Sensitivity and specificity of classification of aTTP | At follow up (180 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the sensitivity and specificity of classification of aTTP patients visits based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Sensitivity and specificity of classification of aTTP | At follow up (365 days) of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  To evaluate the sensitivity and specificity of classification of aTTP patients visits based on HemosIL AcuStar chemiluminescent assay, in comparison with ELISA and/or FRETS.
Clinical characteristics | At diagnosis of patients with acquired thrombotic thrombocytopenic purpura (aTTP).
  Describe clinical characteristics of patients with TMA at the diagnosis and those with aTTP at the diagnosis and follow up based on ADAMTS13 cut-off < 10%.
Clinical characteristics | At follow up (10 days)
  Describe clinical characteristics of patients with TMA at the diagnosis and those with aTTP at the diagnosis and follow up based on ADAMTS13 cut-off < 10%.
Clinical characteristics | At follow up (30 days)
  Describe clinical characteristics of patients with TMA at the diagnosis and those with aTTP at the diagnosis and follow up based on ADAMTS13 cut-off < 10%.
Clinical characteristics | At follow up (60 days)
  Describe clinical characteristics of patients with TMA at the diagnosis and those with aTTP at the diagnosis and follow up based on ADAMTS13 cut-off < 10%.
Clinical characteristics | At follow up (90 days)
  Describe clinical characteristics of patients with TMA at the diagnosis and those with aTTP at the diagnosis and follow up based on ADAMTS13 cut-off < 10%.
Clinical characteristics | At follow up (180 days)
  Describe clinical characteristics of patients with TMA at the diagnosis and those with aTTP at the diagnosis and follow up based on ADAMTS13 cut-off < 10%.
Clinical characteristics | At follow up (365 days)
  Describe clinical characteristics of patients with TMA at the diagnosis and those with aTTP at the diagnosis and follow up based on ADAMTS13 cut-off < 10%.

CONTACTS AND LOCATIONS:
Locations (6):
- Centro Hospitalar e Universitario de Coimbra, Coimbra, Coimbra District, Portugal
- Spain (5):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital La Fe de Valencia, Valencia